CLINICAL TRIAL: NCT06005532
Title: Randomized Double Blind Phase III Trial Comparative Clinical Safety, Efficacy and Immunogenicity of Adalimumab (Manufactured by Mabscale, LLC) to Humira®.
Brief Title: Study Evaluation of the Efficacy, Safety and Immunogenicity of Adalimumab in Comparison With Humira®
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabscale, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MABPS-3/2020
Record Dates: First submitted 2023-07-05; First posted 2023-08-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adalimumab (manufactured by Mabscale, LLC) (Experimental): In the main period, patients will begin Visit 1 receiving Adalimumab therapy at an initial dose (80 /0, 16 ml) on Visit 1, from Visit 2 Adalimumab therapy at a maintenance dose (40 /0, 8 ml) for up to Visit 9 of therapy. Each visit is conducted every two weeks ± 2 days. In additional period (from Visit 11 until Visit 28), eligible patients will continue to receive treatment after additional randomization (Adalimumab or Humira® (40 /0, 8 ml)) every 2 weeks until the end of a trial.
  Interventions: Drug: Adalimumab
- Humira® (Active Comparator): In the main period, patients will begin Visit 1 receiving Humira® therapy at an initial dose (80 /0, 8 ml) on Visit 1, from Visit 2 Humira® therapy at a maintenance dose (40 /0, 4 ml) for up to Visit 9 of therapy. Each visit is conducted every two weeks ± 2 days.
  In additional period (from Visit 11 until Visit 28), eligible patients will continue to receive treatment after additional randomization (Adalimumab or Humira® (40 /0, 4 ml)) every 2 weeks until the end of a trial.
  Interventions: Drug: Humira

INTERVENTIONS:
Drug: Adalimumab — Adalimumab injection 40 mg / 0.8 ml
  Arms: Adalimumab (manufactured by Mabscale, LLC)
Drug: Humira — Adalimumab injection 40 mg / 0.4 ml
  Arms: Humira®

SUMMARY:
MABPS-3/2020 is a double-blind randomized multicenter clinical trial comparing efficacy, immunogenicity and safety profiles of Adalimumab (manufactured by Mabscale, LLC) compared to Humira®.

The purpose of the study is to demonstrate efficacy, immunogenicity and safety of Adalimumab (manufactured by Mabscale, LLC) to Humira ® in adult patients with chronic plaque psoriasis of moderate and severe degree.

DETAILED DESCRIPTION:
Adalimumab is a recombinant humanized monoclonal antibody currently being developed by Mabscale LLC, as a proposed biosimilar to Humira®, which is approved as treatment in patients with chronic plaque psoriasis.

This randomized equivalence study is designed to meet the regulatory requirement for approval of a biosimilar product.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male and female patients aged 18-65 years, body weight ≥ 50 kg and ≤ 120 kg.
3. Established clinical diagnosis plaque psoriasis, lasting at least 6 months before the screening.
4. Plaque psoriasis of moderate or severe severity of stable course with:

   * PASI ≥ 12 points;
   * BSA ≥ 10 %;
   * sPGA ≥ 3 points.
5. Patients who have been shown to undergo systemic therapy and/or patients who have had insufficient therapeutic efficacy of at least 1 previous standard systemic therapy for psoriasis, including phototherapy, therapy with cytostatic and immunosuppressive drugs, or who have had intolerance to standard systemic therapy.

Exclusion Criteria:

1. Data on intolerance or hypersensitivity to any components of the drugs, or to any other human proteins, immunoglobulin preparations.
2. A history of severe hypersensitivity reactions of any etiology.
3. Other (other than plaque) forms of psoriasis.
4. Drug-induced psoriasis.
5. Data on the use of the Adalimumab or any preparations of monoclonal antibodies inhibiting TNF-α at any time during life.
6. The presence of Adalimumab antibodies.
7. Extensive surgical intervention performed less than 30 days before the screening period, or planned extensive surgical intervention during the study period.
8. Active or latent tuberculosis
9. Lymphoproliferative diseases, lymphoma, leukemia, myeloproliferative diseases or a history of multiple myeloma.
10. Any other malignant neoplasms currently or in anamnesis within the last 5 years, with the exception of completely removed and/or cured.
11. Confirmed coronavirus infection caused by COVID-19 within 8 weeks prior to the screening period.
12. Anamnestic data on the presence of syphilis, viral hepatitis B, viral hepatitis C, HIV.
13. Vaccination with live or attenuated vaccines within 8 weeks before the screening period.
14. Hepatic and/or renal insufficiency.
15. Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieved a response according to the PASI criterion of 75 (a decrease in the severity and prevalence of psoriasis by ≥75% from the baseline level assessed by the PASI index) | after 16 weeks of therapy (assessment at Visit 10)
Proportion of patients with positive antibody titer to Adalimumab | 51 weeks of therapy
Percentage of patients who have neutralizing antibodies to Adalimumab | 51 weeks of therapy

CONTACTS AND LOCATIONS:
Locations (9):
- Russia (9):
  - Regional dermatovenerologic dispensary, Barnaul
  - Chelyabinsk Regional Clinical Dermatovenerologic Dispensary, Chelyabinsk
  - Interregional Clinical Diagnostic Center, Kazan'
  - City clinical hospital n.a.Botkin, Moscow
  - Rheumatology research Instititue n.a.Nasonova, Moscow
  - State Scientific Center of Dermatovenerology and Cosmetology, Nizhny Novgorod
  - Reafan, Novosibirsk
  - New Clinic, Pyatigorsk
  - Dermatovenerologic dispensary N10, Saint Petersburg